CLINICAL TRIAL: NCT04990752
Title: Effects of Ulinastatin on Persistent Inflammatory Response During ECMO Support
Brief Title: Effects of Ulinastatin on Inflammatory Response During ECMO Support
Acronym: Uli-ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Huadu District People's Hospital of Guangzhou (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Dongguan People's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-154
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-06

CONDITIONS: ECMO; Inflammatory Response
Keywords: ulinastatin
MeSH Terms: interventions — urinastatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: None Retained — blood sample
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The ulinastatin group: In the ulinastatin group, ulinastatin was used for inflammation management and organ protection early before ECMO was started. The recommended dosage of ulinastatin is 300,000 IU, q8h (Continuous administration for more than 5 days).
  Interventions: Drug: ulinastatin
- The control group: In the control group, patients were treated with conventional treatment without ulinastatin.

INTERVENTIONS:
Drug: ulinastatin — In the ulinastatin group, early application of ulinastatin was performed for inflammation management and organ protection before ECMO initiation.The recommended clinical routine dosage of ulinastatin is 300,000 IU, q8h (continuous administration for more than 5 days).
  Groups: The ulinastatin group

SUMMARY:
This study is a multicenter, prospective, observational cohort study. The subjects were patients who received ECMO support. According to whether ulinastatin is used in the treatment regimen (determined by the competent doctor according to the patient's condition), the patients were divided into the ulinastatin and control groups. In the ulinastatin group, ulinastatin was used for inflammation management and organ protection early before ECMO was started. Baseline data and inflammatory markers (CRP, IL-6, IL-10, TNF-α), capillary leakage markers, routine test results, duration of ECMO use/length of hospital stay/length of ICU stay were recorded at 1, 3, and 5 days after the start of ECMO support, and patients were followed up on the 28th and 90th days.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, observational cohort study. The subjects were patients who received ECMO support. According to whether ulinastatin is used in the treatment regimen (determined by the competent doctor according to the patient's condition), the patients were divided into the ulinastatin and control groups. 144 subjects were enrolled, including 72 subjects in the ulinastatin group and 72 subjects in the control group. In the ulinastatin group, ulinastatin was used for inflammation management and organ protection early before ECMO was started. The recommended clinical routine dosage of ulinastatin is 300,000 IU, q8h (continuous administration for more than 5 days). Baseline data and inflammatory markers (CRP, IL-6, IL-10, TNF-α), capillary leakage markers, routine test results, duration of ECMO use/length of hospital stay/length of ICU stay were recorded at 1, 3, and 5 days after the start of ECMO support, and patients were followed up on the 28th and 90th days.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent;
* ≥18 years old;
* Patients have indications for ECMO support;

Exclusion Criteria:

* Pregnancy or lactation;
* Withdrawal of ECMO or death of the patient within 48 hours of the start of operation;
* Solid-organ or bone marrow transplant recipients;
* Previous history of allergy to ulinastatin or any ingredient or preservative;
* Patients with autoimmune diseases, tumors, or patients receiving high doses of glucocorticoids or immunosuppressant therapy within 2 months;
* Patients judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indications for receiving ECMO support and who, at the clinician's discretion, need ECMO support.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
CRP level | change from admission to 5 days after ECMO support
  The serum levels of CRP
IL-6 level, IL-10 level | change from admission to 5 days after ECMO support
  The serum levels of IL-6 and IL-10
TNF-α level | change from admission to 5 days after ECMO support
  The serum levels of TNF-α

SECONDARY OUTCOMES:
Capillary leakage index | change from admission to 5 days after ECMO support
  CRP(mg/dl)/ALB(g/L)
Renal function | change from admission to 5 days after ECMO support
  The serum levels of creatinine
Liver function | change from admission to 5 days after ECMO support
  The serum levels of ALTand AST
Myocardial injury indexes | change from admission to 5 days after ECMO support
  The serum levels of cTnT and CK-MB
Cardiac function | change from admission to 5 days after ECMO support
  The serum levels of NT-Pro-BNP
Infection | change from admission to 5 days after ECMO support
  The serum levels of PCT
Immunity | change from admission to 5 days after ECMO support
  The serum levels of LYM and WBC
Incidence of new organ insufficiency/failure during ECMO support | during ECMO support
  Incidence of new organ insufficiency/failure during ECMO support
Duration of use of ECMO/length of hospital stay/length of ICU stay | through study completion
  Duration of use of ECMO/length of hospital stay/length of ICU stay
Mortality rate of in-hospital /28d/90d | 90 days after admission
  Mortality rate of in-hospital /28d/90d

CONTACTS AND LOCATIONS:
Overall Officials: Zhongqing Chen, doctor, Study Chair — Nanfang Hosptial of Southern Medical University
Locations (1):
- Nangfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided